CLINICAL TRIAL: NCT07072351
Title: A Phase Ib/II Study of Hypofractionated Radiotherapy Combined With Immunochemotherapy as Conversion Therapy for Locally Advanced Gastroesophageal Junction Adenocarcinoma
Brief Title: Hypofractionated Radiotherapy Combined With Immunochemotherapy for Conversion Treatment of Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yaqin Zhao, Associate Chief Physician, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEJA-ICRT-2025-05
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Hypofractionated Radiotherapy; Immunotherapy; Chemotherapy
Keywords: hypofractionated radiotherapy; immunotherapy; chemotherapy; ORR; conversion therapy; gastroesophageal junction adenocarcinoma
MeSH Terms: interventions — Radiation Dose Hypofractionation; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (HFRT+ICT) (Experimental)
  Interventions: Radiation: hypofractionated radiotherapy; Drug: SOX Chemotherapy; Drug: PD-1 inhibitor
- Control Arm (nICT) (Active Comparator)
  Interventions: Drug: SOX Chemotherapy; Drug: PD-1 inhibitor

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — In Phase Ib, HFRT will be administered at one of three dose levels: 3 Gy × 5 fractions, 4 Gy × 5 fractions, or 5 Gy × 5 fractions. The recommended dose determined in Phase Ib will be used in Phase II (delivered as 5 fractions).
  Other Names: HFRT; LFRT
  Arms: Intervention Arm (HFRT+ICT)
Drug: SOX Chemotherapy — SOX chemotherapy regimen: Oxaliplatin 130 mg/m² administered by intravenous infusion on Day 1; S-1 administered orally for 14 consecutive days followed by a 7-day rest period. The dosage of S-1 is based on body surface area (BSA): 40 mg twice daily for BSA ≤1.5 m², 50 mg twice daily for BSA between 1.5-1.6 m², and 60 mg twice daily for BSA ≥1.6 m². Each cycle is repeated every 3 weeks.
Drug: PD-1 inhibitor — Sintilimab 200 mg administered by intravenous infusion on Day 1 of each 3-week cycle.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of conversion therapy using HFRT combined with ICT in locally advanced or metastatic unresectable GEJA.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether hypofractionated radiotherapy (HFRT) combined with a PD-1 inhibitor (Sintilimab) and chemotherapy based on the SOX regimen is a safe and well-tolerated conversion strategy for patients with locally advanced or metastatic unresectable gastroesophageal junction adenocarcinoma (GEJA), and whether it can improve the objective response rate (ORR) compared to immunochemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Histologically and/or cytologically confirmed diagnosis of locally advanced gastroesophageal junction adenocarcinoma (GEJA), Siewert type I-III, with staging of cT3-4, any N, M0 or cT2 N+, M0, according to the AJCC 8th edition.
2. Resectable locally advanced disease as determined by multidisciplinary team (MDT) assessment.
3. Age ≥18 years, regardless of sex.
4. ECOG performance status of 0 or 1.
5. Estimated life expectancy of ≥3 months.
6. No prior anti-tumor therapy.
7. At least one measurable lesion per RECIST v1.1, defined as:

   * Lesion ≥1 cm in longest diameter on spiral CT, or
   * Lesion ≥2 cm in longest diameter on conventional CT or MRI.
   * Imaging must be performed within 28 days prior to enrollment.
8. Adequate organ function within 14 days prior to treatment, as defined below (Note: No RBC or platelet transfusion or use of G-CSF within 14 days prior to hematology testing):

   Hematologic:
   * Hemoglobin ≥9 g/dL (without transfusion)
   * ANC ≥1.5 × 10⁹/L
   * WBC ≥3.0 × 10⁹/L (without G-CSF)
   * Platelets ≥75 × 10⁹/L (without IL-11 or TPO)

   Biochemical:
   * Total bilirubin ≤1.5 × ULN
   * AST and ALT ≤2.5 × ULN
   * Serum creatinine ≤1.5 × ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault formula)
   * Albumin ≥25 g/L (2.5 g/dL)

   Coagulation (within 7 days prior to enrollment):
   * INR <1.5
   * APTT <1.5 × ULN
   * INR or PT ≤1.5 × ULN
9. For patients with active hepatitis B or C:

   * Antiviral therapy must be initiated ≥14 days before enrollment
   * HBV DNA ≤500 IU/mL or ≤2500 copies/mL; HCV RNA undetectable
   * Must agree to continue antiviral therapy during the study
10. Left ventricular ejection fraction (LVEF) ≥50% by echocardiography.
11. Women of childbearing potential:

    * Negative serum or urine pregnancy test within 7 days prior to enrollment
    * Agree to use effective contraception during the study and for at least 3 months after the last dose
    * Must not breastfeed or donate/retrieve ova within 60 days after the last dose
    * Effective contraception must be continued for at least 6 months after last dose of chemotherapy
12. Men must be surgically sterile or agree to use effective contraception during the study and for at least 3 months after the last dose.
13. Voluntarily signed informed consent with good compliance and willingness to complete study procedures and follow-up.

Exclusion Criteria:

Participants who meet any of the following conditions will be excluded:

1. Diagnosed as mismatch repair deficient (dMMR) or microsatellite instability-high (MSI-H) by immunohistochemistry or gene testing.
2. Evidence of peritoneal or multi-organ metastatic disease, as confirmed by chest and abdominal CT, bone scan, or MRI (in cases with suspected osseous lesions).
3. History of or concurrent other malignancies within the past 5 years, excluding cured basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
4. Known allergy to any component of the investigational drugs, history of severe hypersensitivity, or any contraindication to study drugs.
5. Clinically significant upper gastrointestinal bleeding within 30 days prior to enrollment or randomization.
6. History of congenital pulmonary fibrosis, drug-induced pneumonitis, active pulmonary tuberculosis, or CT-confirmed active pneumonia; interstitial lung disease requiring steroid treatment.
7. Active autoimmune or inflammatory diseases requiring immunosuppressive therapy within 2 years prior to treatment, including but not limited to:

   * Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, diverticulitis),
   * Systemic lupus erythematosus,
   * Sarcoidosis,
   * Tuberculosis,
   * Wegener's granulomatosis,
   * Myasthenia gravis,
   * Graves' disease,
   * Rheumatoid arthritis,
   * Hypophysitis,
   * Uveitis,
   * Glomerulonephritis,
   * Nephrotic syndrome,
   * Fanconi syndrome, or renal tubular acidosis. Exceptions: type 1 diabetes, hypothyroidism controlled by hormone replacement, and non-systemically treated dermatologic conditions (e.g., vitiligo, psoriasis, alopecia).
8. History of immunodeficiency, HIV infection (positive HIV 1/2 antibodies), congenital or acquired immunodeficiency disorders, or history of organ transplantation.
9. Active hepatitis B (HBsAg positive) or active hepatitis C infection. Patients with past or controlled HBV/HCV infection may be eligible.
10. Use of systemic corticosteroids or immunosuppressants within 2 weeks prior to study treatment.

    * Inhaled or topical corticosteroids and adrenal replacement doses (equivalent to ≤10 mg/day prednisone) are permitted.
    * Short-term (<7 days) corticosteroids are allowed for non-autoimmune conditions or prophylaxis (e.g., contrast allergy).
11. Uncontrolled or serious comorbidities, including:

    * Poorly controlled hypertension (SBP ≥150 mmHg or DBP ≥100 mmHg despite medication)
    * Myocardial infarction, ischemia (grade II or above), acute coronary syndrome within 6 months, arrhythmia (e.g., QTc ≥480 ms, atrial fibrillation), or uncontrolled angina
    * NYHA class III-IV heart failure, LVEF <50%, severe valvular disease, cardiomyopathy of any cause
    * History of stroke or transient ischemic attack within screening period
    * Active or uncontrolled infection
    * Severe liver disease (e.g., cirrhosis, decompensated liver disease, chronic active hepatitis) affecting tolerability to treatment
    * Poorly controlled diabetes (fasting glucose >10 mmol/L)
    * Proteinuria ≥++ on dipstick or >1.0 g/24 h on urine protein quantification
12. Coagulation disorders (INR >1.5 or APTT >1.5 × ULN), bleeding tendency, or current use of thrombolytics or anticoagulants.

    * Known hereditary or acquired bleeding/thrombotic conditions (e.g., hemophilia, coagulopathy, thrombocytopenia, hypersplenism).
    * History of significant hemoptysis (≥2.5 mL/day) or massive bleeding within 2 months.
    * Gastrointestinal bleeding, bleeding gastric ulcer, positive fecal occult blood (++ or above), vasculitis, or active bleeding within 3 months.
    * Long-term use of warfarin/heparin or high-dose antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).
13. Major surgery (e.g., craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose, or planned major surgery during the study period.
14. Gastrointestinal perforation and/or fistula within 6 months prior to enrollment; history of arterial/venous thrombotic events such as stroke (excluding clinically stable infarction per investigator), deep vein thrombosis, or pulmonary embolism.
15. Unhealed wounds or fractures of clinical significance.
16. Severe gastrointestinal conditions that may impair oral medication absorption (e.g., dysphagia, chronic diarrhea, intestinal obstruction).
17. Severe malnutrition.
18. Pregnant or breastfeeding women, or subjects (male or female within one year of menopause) unwilling to use effective contraception.
19. History of substance abuse or uncontrolled psychiatric disorders.
20. Unwilling or unable to comply with study procedures.
21. Participation in another interventional clinical trial within 30 days prior to first dose or planning to do so during the current study.
22. Any other condition deemed by the investigator to pose significant risk to patient safety or interfere with study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-05-14 (Estimated); Study Completion 2028-05-14 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability in Phase Ib | within 3 months after the HFRT
  Safety will be assessed based on clinical adverse events, vital signs, and abnormalities in laboratory tests during the study period.
  Adverse events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
  All deaths occurring within 90 days after the first dose of treatment or within 30 days after the last dose will be listed along with the causes of death.
  Laboratory abnormalities will be categorized according to NCI-CTCAE version 5.0.
  Maximum Tolerated Dose (MTD): If ≥1 out of 3 patients in a given dose cohort experiences radiotherapy-related dose-limiting toxicity (DLT) within 90 days, that dose level will be considered intolerable. The next lower dose level will be defined as the MTD. The MTD cohort must include at least 6 evaluable patients.
ORR rate in Phase II | approximately 4 weeks after the resection of primary lesion
  Objective Response Rate (ORR):ORR is defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR) as determined by investigators based on RECIST version 1.1. The initial CR or PR must be confirmed by repeat imaging at least 4 weeks after the first documentation of response.

SECONDARY OUTCOMES:
R0 resection rate | approximately 2 weeks after the resection of primary lesion
  number of R0 surgery divide all participants
DOR (Duration of Response) | Up to 3 years
  Duration from the first documented complete response (CR) or partial response (PR) to the date of disease progression (PD) or death from any cause.
PFS (Progression-Free Survival) | Up to 3 years
  Time from the first administration of the study treatment to disease progression (PD) or death from any cause, whichever occurs first.
OS (Overall Survival) | Up to 3 years
  Time from the initiation of study treatment to death from any cause.
Adverse Events (AEs) | From the first dose through 90 days after the last dose
  The incidence, severity, and relationship of adverse events will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Quality of Life (QoL) - EORTC QLQ-C30 | At baseline, during treatment, and at predefined follow-up visits
  Quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - West China Xiamen Hospital, Sichuan University, Xiamen, Fujian
  - The Seventh People's Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - West China Shangjin Nanfu Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
IPD(individual patient data) Sharing Plan: Shared for: scientific research institutions, academic journal editors, government agencies Sharing conditions: IPD sharing shall meet the following conditions: Requestor must provide study agreement and relevant ethical review committee approval documents Requestor must ensure legality of data use and privacy protection Requestor must agree to data sharing, and the study team has the right to review the Requestor 's study plan and provide necessary support and interpretation of data
  Scope of shared data: The shared data includes ECG and clinical data of all subjects, but excluding personal information of subjects